CLINICAL TRIAL: NCT02807831
Title: A Randomized Clinical Trial Comparing Executive Function and Language Skills Training on School Readiness in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Guilherme Vanoni Polanczyk, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/51.624-1
Record Dates: First submitted 2016-06-10; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Executive Function; Language; Preschool Child
Keywords: Executive Function; Language; Preschool child; Development
MeSH Terms: conditions — Language

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Executive functions training (Experimental)
  Interventions: Behavioral: Executive functions training
- Language skills training (Experimental)
  Interventions: Behavioral: Language skills training
- Regular school curriculum (Active Comparator)
  Interventions: Other: Regular school curriculum

INTERVENTIONS:
Behavioral: Executive functions training — Daily training of executive functions via activities to develop auto-regulation, attention and memory.
  Arms: Executive functions training
Behavioral: Language skills training — Daily training of language skills via activities to develop phonological awareness and vocabulary.
  Arms: Language skills training
Other: Regular school curriculum — Ministry of Education national school curriculum.
  Arms: Regular school curriculum

SUMMARY:
Background: environmental influences in the first years of life have a great impact on adulthood. Adequate environmental stimulation in the first years of life positively influence cognitive, emotional and neurological development. Studies show that high quality education for 3 to 6 years old children are cost-effective for diverse outcomes, such as socioemotional and cognitive development, as well as school performance. However, it is not clear why specific types of interventions are most effective on school readiness, an important precursor of literacy status and later life outcomes. Objectives: adapt to the Brazilian context two well-known intervention programs: (1) executive functions training developed by Diamond, and (2) oral language skills based on the Nuffield Programme developed by Snowling and colleagues. Methods: a randomized controlled trial involving 720 children (4 to 5 years old) allocated to three groups: (1) adapted school curriculum focusing on executive functions training, (2) adapted school curriculum focusing on oral language skills training, and (3) regular school curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Schools interested in the intervention program
* Preschool children (4 to 6 years old)

Exclusion Criteria:

* Presence of any sensory impairment
* Intellectual disability

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 582 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in school readiness | Beginning of the school year (baseline) and at the end of the school year (post intervention, 7 to 8 months later)
  Assessed with a 43 items questionnaire developed by the research staff.

SECONDARY OUTCOMES:
Change in inhibitory control | Beginning of the school year (baseline) and at the end of the school year (post intervention, 7 to 8 months later)
  Inhibitory control assessed via the Flanker e Simon (Dots task) tests.
Change in working memory | Beginning of the school year (baseline) and at the end of the school year (post intervention, 7 to 8 months later)
  Working memory assessed via the neuropsychological Automated Working Memory Assessment (AWMA).
Change in oral language skills | Beginning of the school year (baseline) and at the end of the school year (post intervention, 7 to 8 months later)
  Expressive language assessed via the Child Language Test - ABFW.